CLINICAL TRIAL: NCT00215462
Title: A Phase II Study of Vinorelbine in Unresectable or Metastatic Esophageal and Gastric Adenocarcinoma
Brief Title: Vinorelbine in Unresectable or Metastatic Esophageal and Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Matthew Kulke, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-012
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Esophageal Cancer; Gastric Cancer; Stomach Cancer
Keywords: gastric adenocarcinoma; esophageal adenocarcinoma; vinorelbine
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vinorelbine

SUMMARY:
The purpose of this study is to collect anti-tumor activity of vinorelbine when given to patients with esophageal or gastric tumors. We will also collect information on the toxicities of vinorelbine in these patients.

DETAILED DESCRIPTION:
* Patients will receive vinorelbine intravenously once per week for eight weeks. These treatments will be repeated after the initial eight weeks as long as the patient continues to receive benefit from the treatment. If the patient experiences significant toxicities, the dose may be reduced or the chemotherapy may be discontinued.
* Before beginning treatment and during therapy, routine laboratory tests, scans and x-rays will be done to check the body's response to treatment. A physical exam will be done at the start of the study and before each course of treatment. Scans will be done after eight weeks of therapy.
* Patients will remain on this study as long as their disease does not become worse or they do not experience severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic esophageal adenocarcinoma. Locally unresectable or metastatic gastric adenocarcinoma. Only patients with measurable tumors are eligible.
* No more than one prior chemotherapy regimen
* ECOG performance status of 0-1
* Life expectancy of > 12 weeks
* Greater than or equal to 1,200 calorie/day intake
* ANC > 1,500/mm3
* AST < 3 x ULN
* Total bilirubin < 2.0 ng/dl
* Platelets > 100,000/mm3
* Serum creatinine < 2.0 mg/dl

Exclusion Criteria:

* Prior therapy with vinca alkaloids
* Chemotherapy within the past three weeks
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Peripheral neuropathy > 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2000-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To assess the anti-tumor activity of vinorelbine when administered to patients with locally advanced or metastatic esophageal or gastric adenocarcinoma.

SECONDARY OUTCOMES:
To evaluate the toxicities of vinorelbine in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts